CLINICAL TRIAL: NCT05062564
Title: Evaluation of the Efficacy of LipiFlow Thermal Pulsation Treatment Performed Before Cataract Surgery in Patients Affected by Meibomian Gland Dysfunction in Reducing Postoperative Dry Eye Disease
Brief Title: Efficacy of LipiFlow in Patients Affected by Meibomian Gland Dysfunction in Reducing Post-cataract Surgery Dry Eye
Acronym: LIPICAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Rita Mencucci, Principal Investigator, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19220/SPE
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Meibomian Gland Dysfunction; Cataract; Surgery--Complications; Dry Eye; Blepharitis
MeSH Terms: conditions — Meibomian Gland Dysfunction; Cataract; Dry Eye Syndromes; Blepharitis | interventions — Massage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LipiFlow group (Experimental): Single preoperative treatment with the thermal pulsation system LipiFlow within two months before cataract surgery
  Interventions: Device: LipiFlow Thermal pulsation system
- Control group (Active Comparator): Eyelid warm compresses plus eyelid massage twice a day for the preoperative month
  Interventions: Procedure: Eyelid warm compresses plus massages

INTERVENTIONS:
Device: LipiFlow Thermal pulsation system — Single treatment with LipiFlow thermal pulsation system on the eyelids within two months before surgery
  Arms: LipiFlow group
Procedure: Eyelid warm compresses plus massages — Eyelid warm compresses plus massages twice a day for the preoperative month
  Arms: Control group

SUMMARY:
Dry Eye Disease (DED) is a disease of the ocular surface which may be secondary to a variety of causes, including cataract surgery. DED is characterized by loss of tear film stability and dry eye symptoms, and its pathogenesis is related to corneal nerve injury, decreased goblet cells, inflammation of the ocular surface, and dysfunction of the meibomian glands (MGD). MGD is the main cause of evaporative DED and can cause irregularity of the ocular surface, affecting the accuracy of the biometric calculation. In addition, it is a risk factor for DED exacerbation after cataract surgery, that may occur in about 40% of cases. Current therapies for DED include artificial tears, warm compresses, manual squeezing of the glands, eyelid hygiene, omega-3 fatty acids, topical cyclosporine, serum tears, topical azithromycin, oral doxycycline. The above therapies in some cases can provide only transient relief, affecting the outcome of cataract surgery and the quality of life of patients. Therefore, stabilization of the ocular surface before cataract surgery is important to achieve better post-operative comfort and a better refractive result. The introduction of LipiFlow thermal pulsation treatment (LTP) represents a controlled method of squeezing the obstructed Meibomian glands by applying heat to the upper and lower eyelids and simultaneously applying pulsatile pressure to the eyelid skin surfaces. The aim of our study will be to evaluate the effect of preoperative LipiFlow therapy in patients with age-related cataracts and mild to moderate MGD in reducing postoperative DED.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years old
* Patients affected by age-related cataract <3 according to the Lens Opacities Classification System III scale (LOCS III)
* Meibomian gland dysfunction (MGD) diagnosed using slit lamp examination, following the criteria reported in the paper Arita R. et al, Am J Ophthalmol. 2016 Sep;169:125-137.
* Fluorescein tear BUT <7 seconds

Exclusion Criteria:

* Subjects with documented history and / or clinical signs of concomitant presence of an eye infection caused by viruses such as herpes simplex virus (HSV) or fungi in the previous 3 months.
* Patients with anterior blepharitis or Demodex
* Meibomian gland atrophy score greater than 2/3
* Subject treated with drugs that can have effects on MGD prior to inclusion in the study
* Active ocular inflammation or history of chronic eye inflammation recurrent in the previous 3 months (e.g. retinitis, macular inflammation, choroiditis, uveitis, iritis, scleritis, episcleritis, keratitis)
* Eyelid abnormalities affecting eyelid function (entropion, ectropion, neoplasia, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis)
* Abnormalities of the ocular surface that compromise the integrity of the cornea (e.g.

previous chemical burn, recurrent corneal erosion, corneal epithelial defect, corneal dystrophy)

* Subjects who underwent eye surgery in the previous 3 months, including intraocular, oculo-plastic, corneal or refractive surgery
* Patients suffering from diabetes mellitus, rheumatism, immune diseases and other serious systemic diseases
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
NIBUT (Non-Invasive Break-Up Time) | The difference between the change in NIBUT of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)
  The difference between the change in NIBUT of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)

SECONDARY OUTCOMES:
Tear meniscus height | The difference between the change in tear meniscus height of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)
  The difference between the change in tear meniscus height of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)
Schirmer test I | The difference between the change in Schirmer test I of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)
  The difference between the change in Schirmer test I of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)
Corneal fluorescein staining | The difference between the change in corneal fluorescein staining of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)
  The difference between the change in corneal fluorescein staining of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)
SPEED (Standard Patient Evaluation of Eye Dryness Questionnaire) questionnaire score | The difference between the change in SPEED questionnaire score of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)
  The difference between the change in SPEED questionnaire score of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)
Meibomian gland status assessed using confocal microscopy | The difference between the change in Meibomian gland status of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)
  The difference between the change in Meibomian gland status of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)
Eyelid margin assessed using slit lamp examination | The difference between the change in eyelid margins of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)
  The difference between the change in eyelid margins of LipiFlow group and control group between Visit 0 (screening/baseline) and Visit 2 (one month after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mencucci, MD, Principal Investigator — AOU Careggi
Locations (1):
- Eye clinic, Careggi University hospital, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: No
We have not planned to share individual participant data (IPD)

REFERENCES:
- [Result] Arita R, Minoura I, Morishige N, Shirakawa R, Fukuoka S, Asai K, Goto T, Imanaka T, Nakamura M. Development of Definitive and Reliable Grading Scales for Meibomian Gland Dysfunction. Am J Ophthalmol. 2016 Sep;169:125-137. doi: 10.1016/j.ajo.2016.06.025. Epub 2016 Jun 23. PMID 27345733
- [Derived] Mencucci R, Mercuri S, Cennamo M, Morelli A, Favuzza E. Efficacy of vector thermal pulsation treatment in reducing postcataract surgery dry eye disease in patients affected by meibomian gland dysfunction. J Cataract Refract Surg. 2023 Apr 1;49(4):423-429. doi: 10.1097/j.jcrs.0000000000001124. PMID 36729441